CLINICAL TRIAL: NCT02185937
Title: Influence of an Acidic Beverage (Coca-Cola) on the Exposure to Imatinib (GLIvec) After Major gastrecTomY in Patients With Gastrointestinal Stromal Tumors (ABILITY)
Brief Title: Influence of an Acidic Beverage on the Imatinib Exposure After Major Gastrectomy
Acronym: ABILITY
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: inclusion was too slow
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ABILITY
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal Stromal Tumor; Major Gastrectomy
Keywords: imatinib; gastrectomy; gastrointestinal stromal tumor; pharmacokinetics
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- water (No Intervention): imatinib intake with water
- cola (Active Comparator): imatinib intake with cola
  Interventions: Dietary Supplement: cola

INTERVENTIONS:
Dietary Supplement: cola — imatinib intake with coca-cola
  Other Names: Coca-cola
  Arms: cola

SUMMARY:
The most common sites for GIST to occur are the stomach (60-70%) and proximal small intestines (20-25%). Therefore patients with GIST often have altered GI-tract due to tumor resection or palliative surgery which might affect imatinib exposure. Indeed, Yoo et al. showed that steady state imatinib trough levels in patients with advanced GISTs after major gastrectomy are lower compared to patients with a previous wedge resection or without gastric surgery. Patients that underwent major gastrectomy had an average imatinib plasma trough levels below 1000 µg/L. This while imatinib trough levels above 1000 µg/L are correlated to more beneficial treatment out-comes (longer Progression Free Survival).

Since imatinib easily and rapidly dissolves at pH 5.5 or less, a lack of gastric acid secretion might be causing the decreased exposure in the patients that underwent major gastrectomy.

Therefore the investigators would like to study if the exposure to imatinib in patients after major gastrectomy can be improved by creating a more acidic environment for absorption through combining imatinib intake with Coca-Cola.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patients with GIST, who previously underwent major gastrectomy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
* Already selected to receive imatinib therapy in a dose of 400-800mg imatinib daily, as judged by the treating physician and with respect for and in agreement with the registration guidelines
* Subject is able and willing to sign the Informed Consent Form prior to screening

Exclusion Criteria:

* Concomitant administration of any anti-cancer therapies (e.g. chemo-therapy, other targeted therapy, experimental drug, etc) other than imatinib
* Concomitant use of medication which strongly inhibits or induces CYP3A4
* Refractory nausea and vomiting, malabsorption with other causes than gastrectomy or external biliary shunt that would preclude adequate absorption.
* Unwillingness to use Coca-Cola
* Unwillingness or inability to swallow whole tablets
* Inability to comply with the requirements of the protocol
* Inability to understand the nature and extent of the study and the procedures required
* Participation in a drug study within 60 days prior to the first day of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
imatinib area under the curve | day 7; predose - 10 hours after dosing
  imatinib exposure assessed as area under the curve

SECONDARY OUTCOMES:
number of adverse events | 2 weeks
  number of adverse events will be reported and compared for both treatments

CONTACTS AND LOCATIONS:
Overall Officials: Nielka van Erp, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

REFERENCES:
- [Result] Lubberman FJE, Gelderblom H, Wilmer CM, Kweekel DM, Desar IME, Colbers A, Burger D, van der Graaf WTA, van Erp N. Does a glass of Coke boost the exposure to imatinib in gastrointestinal stromal tumour patients after gastrectomy? Br J Clin Pharmacol. 2017 Oct;83(10):2312-2314. doi: 10.1111/bcp.13333. Epub 2017 Jul 4. No abstract available. PMID 28677263